CLINICAL TRIAL: NCT02223858
Title: Staying Positive: An Intervention to Reduce Osteoarthritis Pain Disparities
Brief Title: Staying Positive With Arthritis Study
Acronym: SPA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Health Services Research
Other Study IDs: IIR 13-080
Record Dates: First submitted 2014-08-18; First posted 2014-08-22 (Estimated); Results first posted 2019-02-11 (Actual); Last update posted 2019-04-03 (Actual); Status verified 2019-03

CONDITIONS: Arthritis
Keywords: Health Status Disparities; Arthritis; Psychology; Pain Management; Affect
MeSH Terms: conditions — Arthritis; Agnosia

STUDY DESIGN:
Intervention Model Description: Randomization will be at the patient level, stratified by study site and patient race, with a 1:1 allocation using random block sizes of 2, 4, 6, or 8.
Who Masked: Participant, Outcomes Assessor
Masking Description: The statistician will seal PA and AC program workbooks in envelopes following the randomization scheme. To blind participants and staff during the baseline assessment, staff will take the next sealed envelope in the sequence to each baseline visit, to be opened after a patient has consented and completed the baseline assessment. The study staff that complete the baseline visits will be unblinded once a participant's envelope is opened; participants will not be told whether they are in the PA or AC program. Staff who conduct the weekly intervention calls in the 6 weeks following the baseline visit will also be unblinded. To maintain blinding for the collection of outcome measures, study staff members who did not complete the baseline visit or any weekly calls during the 6-week program period for a given participant will collect the 1, 3, and 6-month follow-up assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Positive Activities (PA) (Experimental): Positive Activities (PA) Program
  Interventions: Behavioral: Positive Activities (PA) Program
- Attention Control (AC) (Active Comparator): Attention Control (AC) Program
  Interventions: Behavioral: Attention Control (AC) Program

INTERVENTIONS:
Behavioral: Positive Activities (PA) Program — 6-week program of at-home activities (1 per week) that have been shown to increase positivity. Activities were delivered via activity booklets and oral instructions provided during weekly telephone calls from trained interventionists. Interventionist oriented participants to the booklets and reviewed the first activity at the end of an in-person baseline visit. Booklets contained all instructions patients needed to complete the full program. Interventionists also provided support via weekly calls in which they assessed completion of the previous week's activity, reviewed instructions for the next activity, and helped participants trouble-shoot anticipated barriers.
  Arms: Positive Activities (PA)
Behavioral: Attention Control (AC) Program — 6-week program of at-home activities (1 per week) based on affectively neutral activities from control conditions in studies of positive activities interventions. Activities were delivered via activity booklets and oral instructions provided during weekly telephone calls from trained interventionists. Interventionist oriented participants to the booklets and reviewed the first activity at the end of an in-person baseline visit. Booklets contained all instructions patients needed to complete the full program. Interventionists also provided support via weekly calls in which they assessed completion of the previous week's activity, reviewed instructions for the next activity, and helped participants trouble-shoot anticipated barriers.
  Arms: Attention Control (AC)

SUMMARY:
Arthritis is a painful, disabling condition that disproportionately affects African Americans. Existing arthritis treatments yield only small to moderate improvements in pain and are not effective at reducing racial disparities in arthritis pain. According to the biopsychosocial model of pain, there is a need for novel interventions that target psychosocial factors associated with arthritis outcomes and disparities in outcomes. Evidence from the field of psychology suggests that an intervention designed to develop a positive mindset has the potential to improve pain and functioning and reduce racial disparities in patients with arthritis. Interventions to foster a positive mindset have been developed for clinical patient populations but have not yet been fully tested in patients with arthritis or in Veterans, nor have their effects on racial differences in clinical outcomes been examined. This study will address these gaps by testing the impact of an evidence-based positive activities intervention on pain and functioning in African American and White Veterans with knee arthritis.

DETAILED DESCRIPTION:
Background: Arthritis is a prevalent and disabling source of chronic pain for which African Americans (AAs) bear a disproportionate burden. The purpose of this study is to test a patient-centered, non-invasive intervention to improve pain outcomes and reduce disparities in AA and White Veterans with knee arthritis. The intervention is designed to help Veterans develop a positive mindset, the health benefits of which are well-documented.

Objectives: The primary aim of this study is to evaluate the impact of a positive intervention on pain and physical functioning in AA and White Veterans with knee arthritis through a randomized, controlled, clinical trial. It is hypothesized that patients randomized to a positive activities (PA) intervention will experience improved pain and functioning compared to patients randomized to an attention control (AC) program, and that these improvements will be larger for AA than for WH Veterans. The secondary aim of this study is to identify variables that mediate the effects of the PA intervention on pain and functioning. It is hypothesized that the effects of the PA intervention will be mediated by psychosocial variables known to be associated with arthritis outcomes or racial differences in arthritis outcomes (e.g., depression, self-efficacy, pain coping, perceived discrimination).

Methods: A randomized, controlled, 2-arm design will be used to compare the effects of a 6-week PA intervention with that of an AC program on pain and functioning at 1, 3, and 6-months post-intervention among AA and WH Veterans with knee arthritis. Approximately 180 AA and 180 WH primary care patients with knee pain symptoms consistent with arthritis will be recruited from participating VA medical centers following the original protocol. [Due to accelerated recruitment of the original target sample, up to 240 additional primary care patients with knee pain symptoms consistent with OA will be recruited from participating VA medical centers using inclusion criteria that take into account original ICD-9 codes and their corresponding ICD-10 codes. The additional patients (including some men and some women, as resources allow) will be recruited to increase power to detect sex differences in secondary analyses after the primary aims of the study have been achieved using the original cohort.] Eligible participants will complete an in-person baseline assessment of study outcomes, mediators, and control variables and be randomized to a 6-week PA or AC program. The PA program consists of completing 6 at-home activities (1 per week) that have been shown to increase positivity. The AC program consists of 6 affectively neutral activities. Both groups will receive weekly telephone calls from trained interventionists to clarify instructions for the next week's activity and assess completion of the previous week's activity. Outcomes and proposed mediating variables will be assessed via telephone surveys at 1 month, 3 months, and 6 months post-intervention. Study outcomes include self-reported pain and physical functioning as measured by the Western Ontario MacMaster Index. Hypothesized mediators include depressive symptoms, positive/negative affect, satisfaction with life, arthritis self-efficacy, pain coping, pain catastrophizing, perceived discrimination, global stress, and social support. The intervention impact over time and by race (primary aim) will be tested using linear mixed models that allow repeated measures on the continuous outcomes for each participant and assess change in outcomes over time. A multiple mediator bootstrap approach to assess whether the effect of the intervention is mediated by the hypothesized mediators.

ELIGIBILITY:
Inclusion Criteria:

The target population will be African American (AA) and White (WH) Veterans with symptomatic knee arthritis. Specific inclusion criteria include:

* Age 50 years or older
* Receive primary care at a participating study site
* Self-report as non-Hispanic black/AA or non-Hispanic WH
* Frequent, symptomatic knee pain identified using questions from the OA Initiative
* Pain level of 4 or higher on a 0-10 numeric rating scale
* Can speak, read, and write in English

Exclusion Criteria:

Patients will be excluded if they:

* Report serious problems with hearing, eyesight, or memory
* Report having been diagnosed any type of arthritis other than osteoarthritis or degenerative arthritis
* Report that they have been treated for cancer in the last 3 years
* Report having had a steroid injection into one or both knees in the past 3 months
* Report having had a knee replacement into one or both knees in the past 3 months
* Report having plans to have a knee replacement in one or both knees in the next 6 months
* Report that there is a reason they cannot complete the study procedures, which include telephone calls and program activities that involve reading and writing
* Do not have a telephone number where they can receive telephone calls from research staff
* Screen positive for cognitive impairment

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2015-07-13 (Actual); Primary Completion 2017-11-09 (Actual); Study Completion 2017-11-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leslie RM Hausmann, PhD, Principal Investigator — VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA
Locations (2):
- United States (2):
  - Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA, Philadelphia, Pennsylvania
  - VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hausmann LRM, Ibrahim SA, Kwoh CK, Youk A, Obrosky DS, Weiner DK, Vina E, Gallagher RM, Mauro GT, Parks A. Rationale and design of the Staying Positive with Arthritis (SPA) Study: A randomized controlled trial testing the impact of a positive psychology intervention on racial disparities in pain. Contemp Clin Trials. 2018 Jan;64:243-253. doi: 10.1016/j.cct.2017.09.001. Epub 2017 Sep 8. PMID 28893676
- [Background] Hausmann LRM, Youk A, Kwoh CK, Ibrahim SA, Hannon MJ, Weiner DK, Gallagher RM, Parks A. Testing a Positive Psychological Intervention for Osteoarthritis. Pain Med. 2017 Oct 1;18(10):1908-1920. doi: 10.1093/pm/pnx141. PMID 29044408
- [Result] Vina ER, Hausmann LRM, Obrosky DS, Youk A, Ibrahim SA, Weiner DK, Gallagher RM, Kwoh CK. Social & psychological factors associated with oral analgesic use in knee osteoarthritis management. Osteoarthritis Cartilage. 2019 Jul;27(7):1018-1025. doi: 10.1016/j.joca.2019.01.010. Epub 2019 Feb 1. PMID 30716537
- [Derived] McClendon J, Essien UR, Youk A, Ibrahim SA, Vina E, Kwoh CK, Hausmann LRM. Cumulative Disadvantage and Disparities in Depression and Pain Among Veterans With Osteoarthritis: The Role of Perceived Discrimination. Arthritis Care Res (Hoboken). 2021 Jan;73(1):11-17. doi: 10.1002/acr.24481. PMID 33026710
- [Derived] Hausmann LRM, Youk A, Kwoh CK, Gallagher RM, Weiner DK, Vina ER, Obrosky DS, Mauro GT, McInnes S, Ibrahim SA. Effect of a Positive Psychological Intervention on Pain and Functional Difficulty Among Adults With Osteoarthritis: A Randomized Clinical Trial. JAMA Netw Open. 2018 Sep 7;1(5):e182533. doi: 10.1001/jamanetworkopen.2018.2533. PMID 30646170

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with symptomatic knee OA from Veterans Affairs (VA) medical centers in Pittsburgh and Philadelphia, Pennsylvania, were recruited by mail and telephone. Mailings were sent to patients meeting basic eligibility criteria based on their VA medical records Recruitment for the study ran from July 2015 to February 2017.
Pre-assignment Details: Eligible patients attended an in-person baseline visit where they provided written informed consent, completed a staff-administered baseline assessment, and were randomized to a 6-week positive psychological intervention or neutral control program.
Groups:
- Positive Activities (PA): Positive Activities (PA) Program: PA activities were delivered using a combination of activity booklets and oral instructions provided during weekly telephone calls from trained interventionists. The booklet contains all instructions patients need to complete the full program. The intervention was an individually-based program in which participants completed one new positive psychological activity for the first 5 weeks and repeated their favorite in week 6. Activities, which were adapted for the target population, included recalling and reflecting on positive events; writing a letter of gratitude; cultivating mindfulness; practicing kindness; and increasing engagement in activities that they enjoy, give them a sense of achievement, or bring them closer to others (a variant of behavioral activation).
- Attention Control (AC): Attention Control (AC) Program: AC activities were delivered using a combination of activity booklets and oral instructions provided during weekly telephone calls from trained interventionists. The booklet contains all instructions patients need to complete the full program. The 6-week program consisting of at-home activities (1 completed per week) are based on affectively neutral activities from control conditions in prior studies of positive activities interventions. The control program was identical to the intervention in terms of framing, reading level, format, duration, and delivery, but contained neutral control activities adapted from previous positive psychological intervention studies. Control activities asked participants to recall events that affected them each day, identify ways they could change their life circumstances, recall early memories, record things they did in the past week, plan their day, and repeat their favorite activity in week 6.
Period: Overall Study
Arm/Group | Positive Activities (PA) | Attention Control (AC)
Started | 180 | 180
1-month Follow-up | 156 | 150
3-month Follow-up | 155 | 154
6-month Follow-up | 156 | 154
Completed | 156 | 154
Not Completed | 24 | 26
Not completed — Death | 1 | 1
Not completed — Lost to Follow-up | 6 | 11
Not completed — Withdrawal by Subject | 8 | 5
Not completed — Refused | 9 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Positive Activities (PA) | Attention Control (AC) | Total
Number analyzed (Participants) | 180 | 180 | 360
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 95 | 100 | 195
  >=65 years | 85 | 80 | 165
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 41 | 85
  Male | 136 | 139 | 275
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 180 | 180 | 360
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 90 | 90 | 180
  White | 90 | 90 | 180
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 180 | 180 | 360
Self-reported pain, physical functioning, and global assessment of pain at baseline [Mean (Standard Deviation); unit: units on a scale] — Population: For Pain and Physical Functioning, those who skipped >20% of items within a scale (>1 or >3 items, respectively) were excluded.
  *WOMAC score range: 0-100; higher=worse symptoms. Global assessment was measured by participants considering their knee arthritis pain condition over the past week (0-10; higher=worse pain).
  units on a scale
    Pain (Western Ontario McMaster Index;100=worst)*: number analyzed (Participants) | 179 | 178 | 357
    Pain (Western Ontario McMaster Index;100=worst)* | 50.24 (16.95) | 47.42 (18.07) | 48.83 (17.55)
    Physical functioning (WOMAC; 100=worst)*: number analyzed (Participants) | 177 | 174 | 351
    Physical functioning (WOMAC; 100=worst)* | 47.94 (17.73) | 45.70 (18.53) | 46.82 (18.14)
    Global assessment (0-10; higher=worse)* | 5.13 (2.14) | 4.89 (1.96) | 5.01 (2.06)

OUTCOME MEASURES:

1. Primary Outcome: Self-reported Pain From Baseline to 1, 3, and 6 Months Post-intervention
Description: Pain subscale of the Western Ontario McMaster (WOMAC) Index. Pain is on a scale of 0-100; higher scores mean worse pain.
Time Frame: Baseline to 6 months post-intervention
Population: Participants had the option to skip any questions they did not wish to answer. This explains why the number analyzed in the rows below differs overall number analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Positive Activities (PA) | Attention Control (AC)
Number analyzed (Participants) | 180 | 180
units on a scale
  Baseline: number analyzed (Participants) | 179 | 178
  Baseline | 50.24 (16.95) | 47.42 (18.07)
  1 month: number analyzed (Participants) | 156 | 149
  1 month | 45.42 (18.58) | 43.57 (20.93)
  3 month: number analyzed (Participants) | 155 | 153
  3 month | 43.87 (19.16) | 43.32 (19.13)
  6 month: number analyzed (Participants) | 156 | 153
  6 month | 43.22 (20.97) | 41.59 (19.87)
Statistical Analysis 1: Comparison: Positive Activities (PA) vs Attention Control (AC); Test type: Superiority — A sample size of 360 patients (180 non-Hispanic white and 180 non-Hispanic African American) was chosen based on a priori power calculations to detect a 3-way interaction between treatment group, race, and time, assuming a 20% change in baseline, the WOMAC pain subscales, and a 80% power; p = 0.791, Mixed Models Analysis; All models adjusted for site

2. Primary Outcome: Self-reported Physical Functioning From Baseline to 1, 3, and 6 Months Post-intervention
Description: Difficulty with physical functioning subscale of the Western Ontario McMaster (WOMAC) Index. Physical functioning is on a scale of 0-100; higher scores mean worse physical functioning.
Time Frame: Baseline to 6 months post-intervention
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Positive Activities (PA) | Attention Control (AC)
Number analyzed (Participants) | 180 | 180
units on a scale
  Baseline: number analyzed (Participants) | 177 | 174
  Baseline | 47.94 (17.73) | 45.70 (18.53)
  1 month: number analyzed (Participants) | 156 | 142
  1 month | 44.61 (19.81) | 43.08 (20.97)
  3 month: number analyzed (Participants) | 153 | 147
  3 month | 43.39 (19.01) | 43.32 (19.80)
  6 month: number analyzed (Participants) | 152 | 148
  6 month | 43.89 (20.02) | 41.91 (20.00)
Statistical Analysis 1: Comparison: Positive Activities (PA) vs Attention Control (AC); Test type: Superiority — A sample size of 360 (180 non-Hispanic white and 180 non-Hispanic African American) was chosen based on a priori power calculations to detect a 3-way interaction between treatment group, race, and time, assuming a 20% change in baseline, the WOMAC pain subscales, and a 80% power; p = 0.880, Mixed Models Analysis; All models adjusted for site

3. Other Pre Specified Outcome: Patient Global Assessment of Pain From Baseline to 1, 3, and 6 Months Post-intervention
Description: Self-reported global assessment of pain in the last week using a numeric rating scale. Global assessment of pain is on a scale of 0-10; higher scores mean worse pain.
Time Frame: Baseline to 6 months post-intervention
Population: Participants had the option to skip any questions they did not wish to answer. This explains why the number analyzed in the rows below differs from the overall number analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Positive Activities (PA) | Attention Control (AC)
Number analyzed (Participants) | 180 | 180
units on a scale
  Baseline | 5.13 (2.14) | 4.89 (1.96)
  1 month: number analyzed (Participants) | 156 | 150
  1 month | 4.77 (2.16) | 4.71 (2.21)
  3 month: number analyzed (Participants) | 155 | 154
  3 month | 4.83 (2.10) | 4.69 (2.06)
  6 month: number analyzed (Participants) | 155 | 153
  6 month | 4.82 (2.27) | 4.60 (2.24)
Statistical Analysis 1: Comparison: Positive Activities (PA) vs Attention Control (AC); Test type: Superiority — A sample size of 360 (180 non-Hispanic white and 180 non-Hispanic African American) was chosen based on a priori power calculations to detect a 3-way interaction between treatment group, race, and time, assuming a 20% change in baseline, the WOMAC pain subscale, and a 80% power; p = 0.901, Mixed Models Analysis; All models adjusted for site

ADVERSE EVENTS:
Time Frame: From baseline through 6-months post intervention.
Description: All adverse events that occurred with the participants fell under the definition of "serious adverse events" as they were all hospitalizations. There are no "other (not including serious) adverse events" to report.
Arm/Group | Positive Activities (PA) | Attention Control (AC)
All-Cause Mortality (participants affected / at risk) | 1/180 | 1/180
Serious Adverse Events (participants affected / at risk) | 12/180 | 8/180
Other Adverse Events (participants affected / at risk) | 0/180 | 0/180
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Positive Activities (PA) (N=180) | Attention Control (AC) (N=180)
Hospitalizations unrelated to the study (General disorders) | 4 (4) | 1 (1)
Hospitalizations unrelated to the study (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hospitalizations unrelated to the study (Cardiac disorders) | 3 (3) | 2 (2)
Hospitalizations unrelated to the study (Gastrointestinal disorders) | 3 (3) | 0 (0)
Hospitalizations unrelated to the study (Psychiatric disorders) | 0 (0) | 1 (1)
Hospitalizations unrelated to the study (Renal and urinary disorders) | 0 (0) | 1 (1)
Hospitalizations unrelated to the study (Vascular disorders) | 1 (1) | 0 (0)
Hospitalizations unrelated to the study (Endocrine disorders) | 0 (0) | 1 (1)
Hospitalizations unrelated to the study (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hospitalizations unrelated to the study (Surgical and medical procedures) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Included patients with knee osteoarthritis from 2 VA medical centers; did not assess pain conditions other than arthritis; adherence and outcomes were self-reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-05-18): https://cdn.clinicaltrials.gov/large-docs/58/NCT02223858/Prot_SAP_000.pdf
  • Informed Consent Form (2016-05-18): https://cdn.clinicaltrials.gov/large-docs/58/NCT02223858/ICF_001.pdf